CLINICAL TRIAL: NCT03196843
Title: Radiotherapy Combine With Raltitrexed Versus Radiotherapy Alone in Older Patients With Head and Neck Squamous Cell Carcinoma: a Prospective Randomized Controlled Trial
Brief Title: Radiotherapy Combine With Raltitrexed Versus Radiotherapy Alone in Older Patients With HNSCC.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Lv Xiupeng, Professor, The First Affiliated Hospital of Dalian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCKY2016-65
Record Dates: First submitted 2017-06-11; First posted 2017-06-23 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: raltitrexed; radiotherapy; older patient; head and neck squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — raltitrexed; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Raltitrexed plus Radiation (Experimental): Raltitrexed 2.5mg/m2, iv, every 3 weeks, concurrently with intensity modulated radiotherapy(IMRT)
  Interventions: Drug: Raltitrexed; Radiation: Intensity Modulated Radiotherapy
- Radiation (Active Comparator): Intensity modulated radiotherapy(IMRT) alone radical radiotherapy:70Gy/2Gy/7 weeks preoperative and postoperative adjuvant radiotherapy:50-60Gy/2Gy/5-6 weeks
  Interventions: Radiation: Intensity Modulated Radiotherapy

INTERVENTIONS:
Drug: Raltitrexed — Raltitrexed 2.5mg/m2 on day 1,22,43 during radiotherapy
  Arms: Raltitrexed plus Radiation
Radiation: Intensity Modulated Radiotherapy — Radical radiotherapy:70Gy/2Gy/7 weeks Preoperative and postoperative adjuvant radiotherapy:50-60Gy/2Gy/5-6 week

SUMMARY:
The purpose of this study is to evaluate the efficacy of radiotherapy combine with raltitrexed in older patients with head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
Radiotherapy play a critical role in the treatment of head and neck squamous cell carcinoma. Concurrent chemoradiotherapy can increased patients' survival rate. Most of head and neck squamous cell carcinoma patients are in the age range from 60 to 80 years old. Head and neck cancer begin in concealed anatomic sites that make it difficult to found the disease. Therefore, a larger proportion of patients diagnosed with cancer at a late stage.The tissues of head and neck are closely related to important functions such as respiratory, swallowing. Therefore patients are often accompanied by poor nutritional status, cardiac dysfunction and other chronic diseases.Since the tumor is extensive and it cannot be completely resected.These patients are not suitable for surgery alone. Radical radiotherapy or adjuvant radiotherapy is often administered. In order to increase the treatment efficacy, patients with high risk are commonly treated with concurrent chemoradiotherapy. Concurrent chemoradiotherapy often cause serious side effects. For older patients who often have chronic health conditions or poor ECOG(Eastern Cooperative Oncology Group) score are difficult to tolerate.It is crucial to enhance the efficacy of treatment of head and neck squamous cell carcinoma in older patients without causing significant side effect.

Raltitrexed is a direct and specific thymidylate synthase (TS) inhibitor and it is an alternative option for patients unsuitable for cisplatin based chemoradiotherapy. It is more suitable for the treatment of head and neck squamous cell carcinoma in older patients. It is deserved to further investigation. Researches indicated that raltitrexed has shown efficacy and good safety profile in the treatment of colorectal cancer.

It is rarely reported that intensity modulated radiotherapy plus raltitrexed in the treatment of patients with head and neck squamous cell carcinoma,particularly in older patients.The aim of this study was to compare the efficacy of intensity modulated radiotherapy plus raltitrexed with intensity modulated radiotherapy alone in older patients with squamous cell carcinoma of the head and neck.

According to EORTC(European Organization for Research on Treatment of Cancer)22931 study, The 2-year PFS(progression-free survival) was 48% with chemotherapy alone in squamous cell carcinoma of the head and neck. Planting A et al studied raltitrexed at escalating doses combine with radiotherapy in locally advanced head and neck cancer. The results showed that 12 out of 17 patients remained free of locoregional recurrence after a median follow-up of 24(+) months (range 3-60+ months).The study was designed to detect a 15-20% clinic benefit for patients, using α of 0.05 and a β of 0.20. To achieve this, the number of patients required was 101 per group, according to drup-out rate 10%.

ELIGIBILITY:
Inclusion Criteria:

1. Before participate in the study, patients must understand the treatment plan and willing to participate in the study. Patients must have signed an approved informed consent.
2. Histopathologic confirmed squamous cell carcinoma of head and neck ,including oral cavity, oropharynx, larynx, or hypopharynx.
3. Ages≥65 years,Not limited to gender.
4. ECOG performance status ≤2.
5. Patients with surgical contraindication or reject to surgery.
6. Postoperative TNM(primary tumor,regional nodes,metastasis) staging III~IV, positive surgical margin.
7. without evidence of distant metastases.
8. No contraindication to chemoradiotherapy.
9. Life expectancy > 3 months.
10. Available Organ function: white blood cell≥3.5×109/L, Neutrophils ≥1.5×109/L, Hemoglobin ≥80g/L, Blood platelet>100×109/L; Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST)≤ 2.5 upper limit of normal(ULN); Total bilirubin (TBIL) <1.5 ULN;serum creatinine≤1.5 ULN; creatinine clearance of ≥ 50ml/min

Exclusion Criteria:

1. Patients with a history of any other malignancy.
2. Concomitant treatment with any other anticancer therapy.
3. Patient have contraindication to chemotherapy(eg.uncontrolled coronarism and heart failure; History of myocardial infarction within the past 6 months, Chronic obstructive pulmonary, uncontrolled epileptic attack and other disease that investigator consider it unsuitable for the chemotherapy)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
PFS，Progress Free Survival | 2 years
  Progress free survival defined as time from the first day of treatment until disease progress or death

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 2 years
  Treatment-Emergent Adverse Event is defined according to CTCAE(Common Terminology Criteria for Adverse Events) v.4.0. All the adverse reactions and serious adverse reactions will be recorded based on laboratory tests, physical examination, ECOG performance status, electrocardiogram and etc. And then will be graded according to CTCAE v.4.0.
OS，Overall Survival | 2 years
  Overall survival was defined as time from diagnosis until either death as a result of any cause. For patients who loss to follow-up before death, defined the last follow-up time as the death time
DCR，Disease Control Rate | 2 years
  according to RECIST criterion, defined as CR(complete response) + PR(partial reponse) + SD(stable disease)

CONTACTS AND LOCATIONS:
Locations (1):
- Lv Xiupeng, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No